CLINICAL TRIAL: NCT04177134
Title: French Register of Patients With Spinal Muscular Atrophy
Acronym: SMA
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP190245; N° IDRCB: 2019-A01161-56 (Other: ANSM)
Record Dates: First submitted 2019-09-26; First posted 2019-11-26 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: Spinal Muscular Atrophy
Keywords: spinal muscular atrophy
MeSH Terms: conditions — Muscular Atrophy, Spinal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 9 Years
Biospecimen Retention: Samples Without DNA — Blood sampling for biomarkers, with DNA.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary objectives of the study are to obtain clinically meaningful data on survival and outcomes of all the patients with spinal muscular atrophy (SMA) 5q types 1 through 4 (according to international classification), being followed in the reference centers of the disease in France between September 1, 2016 and August 31, 2024. The registry will collect retrospectively and prospectively the longitudinal data of the long-term follow-up for child and adult patients, under real life conditions of current medical practice, in order to document the clinical evolution of patients (survival, motor, respiratory, orthopedic and nutritional), the conditions of use of the treatments, the mortality rates of treated and untreated patients, the tolerance of the treatments, adverse events in order to better define their places in the therapeutic strategy.

DETAILED DESCRIPTION:
As secondary objectives, the study aims:

* to estimate the frequencies of patients with SMA 5q types 1 through 4 who have being treated in the reference centers between September 1 2016 and August 31 2024;
* to describe overall demographic, familial, clinical, biological, and genetic characteristics of SMA 5q patients treated in all regions of France, by the type of SMA (type 1,2,3, and 4);
* to study the impact of proactive and symptomatic medical interventions (bracing, IPPB devices) and medications (vaccinations, anti-infectious, digestive, nutritional supplements) in the evolution of patients;
* to study the long-term evolution (survival, motor and respiratory functions, spinal shape, growth and nutritional function) of SMA 5q in treated and untreated populations, by new available therapies, throughout the register;
* to study mortality rate of SMA 5q in treated and untreated populations, by new available therapies, throughout the register;
* to identify and document the different therapeutic strategies by sub-populations and by discontinuation or follow-up of treatments;
* to evaluate prognostic factors of responses to therapies;
* to study the tolerance of treatments by type of treatments, by type of SMA and overall tolerance (including adverse events);
* to estimate the costs of care for SMA 5q patients in different groups (types, ages);
* to provide needful elements to evaluate the health care costs for the disease;
* to study the autonomy and the quality of life of patients depending on different therapeutic strategies;
* to study the impact of the disease on caregivers;
* to facilitate development of scientific research on SMA in the conduct of trials on new therapeutic strategies.

ELIGIBILITY:
Inclusion Criteria:

* Genetically confirmed SMA 5q patients through 1 to 4 types treated in reference centers in France between September 1, 2016 and August 31, 2024.
* for prospective study: inform consent form signed by patient.
* for retrospective data: information form with non-opposition have been given to participant.
* Covered by a health insurance.

Exclusion Criteria:

* Other type of SMA (not 5q).
* Under guardianship or curatorship.
* Unable to understand french language.

Min Age: 0 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 1000 SMA 5q patients of type 1, 2, 3 and 4, followed or diagnosed between September 1, 2016 and August 31, 2024. It is estimated that approximately 50% of patients will be children.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-01-31 (Actual); Primary Completion 2029-01-31 (Estimated); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
Motor functional development or status | baseline, 1 year, 2 year, 3 year, 4 year, 5 year, 6 year, 7 year, 8 year and 9 year
  * SMA Type 1 until 2 years of age: change of HINE (Hammersmith Infant Neurological Examination) score
  * Children: change in Vignos and Brooke scores (level of upper and Lower extremities autonomy)
  * Adults: change in Walton & Boston scores (level of upper and Lower extremities autonomy)
Motor function scores | baseline, 1 year, 2 year, 3 year, 4 year, 5 year, 6 year, 7 year, 8 year and 9 year
  * For children ≤ 2 years: change of CHOP INTEND (Children's Hospital of Philadelphia Infant Test of Neuromuscular Disorders) score will be evaluated
  * For children between 2 and 5 years, ambulatory or not: Change of total MFM-20 (Motor Function Measure 20) score will be evaluated. Change of 3 dimension scores will be evaluated: D1 (start and transfers station), D2 (axial and proximal motricity) and D3 (distal including the upper limb)
  * For children children > 6 years and adults, ambulatory or not: Change of total MFM-32 (Motor Function Measure 32) score will be evaluated. Change of 3 dimension scores will be evaluated: D1 (start and transfers station), D2 (axial and proximal motricity) and D3 (distal including the upper limb).
  * For ambulatory individuals: added 6MWT (6 minutes walking test)
Yearly changes of morbi-mortality-vital events | 9 years
  Events of hospitalizations, recurrent infections, fractures, complications and death.
Respiratory events | baseline, 1 year, 2 year, 3 year, 4 year, 5 year, 6 year, 7 year, 8 year and 9 year
  Onset of respiratory support or change in the mode and time (including intubations).
Digestive-nutritional events | baseline, 1 year, 2 year, 3 year, 4 year, 5 year, 6 year, 7 year, 8 year and 9 year
  Digestive events, onset of nutritional support or change in the mode and time
Yearly changes of spinal events | 9 years
  Onset of spinal deformity, or increment of 5° or more in the Cobb angle (examination in supine position without brace ; if sitting possible, examination in the upright position, with or without brace or with or without implant (surgery)

SECONDARY OUTCOMES:
Frequency | through study completion, an average of 9 year
  Frequencies of patients with SMA 5q of type 1,2,3 and 4 cared in the reference centres between September 1 2016 and August 31 2024.
Responses to the treatments (nusinersen and salbutamol) | 1 year, 2 year, 3 year, 4 year, 5 year, 6 year, 7 year, 8 year and 9 year
  Responses of the primary outcome measures to the therapies (salbutamol, nusinersen, onasemnogene, risdiplam)
Spinal status | 1 year, 2 year, 3 year, 4 year, 5 year, 6 year, 7 year, 8 year and 9 year
  Evolution of scoliosis (Cobb angle) in the preoperative period (patients treated vs not treated with Garches brace): first and last Cobb angle (and ages)
Impact of spinal surgery techniques in scoliosis | 1 year, 2 year, 3 year, 4 year, 5 year, 6 year, 7 year, 8 year and 9 year
  Impact of spinal surgery techniques in scoliosis (presurgical and last post surgical Cobb angle)
Mortality | at 1, 2 and 5 years
  For treated and untreated patients. Rate of mortality will be assessed at 1,2 and 5 years.
Pulmonary function | at 6 months
  Forced vital capacity (FVC) will be evaluated at least once per year for children > 5 years, by specifying the posture of realization of the test, lying vs sitting.
Respiratory muscles performance | at 6 months
  Peak expiratory and inspiratory pressures will be evaluated if possible for children > 5 years (MEP, MIP, PF, SNIP (sniff nasal inspiratory pressure)
Pulmonary function | at 6 months
  PCF (peak cough flow) will be evaluated at least once per year for children > 5 years, by specifying the posture of realization of the test, lying vs sitting.
Cardiological parameter | through study completion, an average of 9 year
  ECG abnormality will be evaluated by Holter ECG 24h: P Wave, QRS Complex, QT Interval
Cardiological function and anatomy | through study completion, an average of 9 year
  Anatomic abnormalities will be evaluated by echocardiography.
Biomarkers | baseline, 1 year, 2 year, 3 year, 4 year, 5 year, 6 year, 7 year, 8 year and 9 year
  Change of biomarkers: Neurofilaments and CPK
Patient's quality of life: PedsQL (Pediatric Quality of Life Inventory) Child report | baseline, 1 year, 2 year, 3 year, 4 year, 5 year, 6 year, 7 year, 8 year and 9 year
  Questionary as the "PedsQL Child report" will be used to evaluate patient's quality of life. Total Scale Score: 0.88 Child Self-Report; 0.90 Parent Proxy-Report.
Patient's quality of life: PedsQL parent report concerning child | baseline, 1 year, 2 year, 3 year, 4 year, 5 year, 6 year, 7 year, 8 year and 9 year
  Questionary as the "PedsQL parent report concerning child" will be used to evaluate patient's quality of life. Total Scale Score: 0.88 Child Self-Report; 0.90 Parent Proxy-Report.
Patient's quality of life: QoL-gNMD for adult | baseline, 1 year, 2 year, 3 year, 4 year, 5 year, 6 year, 7 year, 8 year and 9 year
  Questionary as "QoL-gNMD for adult" (Quality of Life in genetic Neuromuscular Disease) will be used to evaluate patient's quality of life.
Caregiver burden assessement | at baseline, 1 year, 2 year, 3 year, 4 year, 5 year, 6 year, 7 year, 8 year and 9 year
  Questionnaire as "Work Productivity and Activity Impairment Questionnaire SMAv2" will be completed once a year by a member of neuromuscular center or patients or their relatives.
Caregiver burden assessement | at baseline, 1 year, 2 year, 3 year, 4 year, 5 year, 6 year, 7 year, 8 year and 9 year
  Questionnaire as "FICD+4 Burden Interview Questionnaire" will be completed once a year by a member of neuromuscular center or patients or their relatives.
  FICD (Family Impact of Childhood Disability)+4 Burden Interview Questionnaire: the multidimensional measurements to assess the impacts on time, expenses, work, relationships and health of caregiver.

CONTACTS AND LOCATIONS:
Overall Officials: Susana Quijano-Roy, MD, PhD, Principal Investigator — Unité neuromusculaire, Service de Neurologie et Réanimation Pédiatrique, Hôpital Raymond Poincaré, 92380 Garches, FRANCE
Locations (1):
- Unité neuromusculaire, Service de Neurologie et Réanimation Pédiatrique, (French neuromuscular reference network (FILNEMUS), Hôpital Raymond Poincaré,, Garches, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Grimaldi L, Garcia-Uzquiano R, de la Banda MG, Oulhissane-Omar A, Tard C, Saugier-Veber P, Laugel V, Desguerre I, Cintas P, Vuillerot C, Audic F, Cances C, Stojkovic T, Urtizberea JA, Attarian S, Ropars J, Quijano-Roy S; Registre SMA France Study Group. REGISTRE SMA FRANCE: A nationwide observational registry of patients with spinal muscular atrophy in France. J Neuromuscul Dis. 2025 Nov;12(6):793-803. doi: 10.1177/22143602251353446. Epub 2025 Jul 8. PMID 40625130
- [Derived] Gerin L, Ropars J, Garcia-Uzquiano R, Gomez-Garcia De la Banda M, Saugier-Veber P, Desguerre I, Salort-Campana E, Espil C, Barnerias C, Laugel V, Cances C, Audic F, Cintas P, Le Goff L, Mallaret M, Nougues MC, Drunat S, Tard C, Grimaldi L, Quijano-Roy S; R-SMA Study Group (FILNEMUS). Spectrum of Phenotypes in SMA Patients With 4 SMN2 Copies in the French Population: Registre SMA France. Neurol Genet. 2025 Apr 1;11(2):e200222. doi: 10.1212/NXG.0000000000200222. eCollection 2025 Apr. PMID 40212804